CLINICAL TRIAL: NCT06379282
Title: Investigating the Role of Energy Balance Modification on Health Responses in Chronic Lymphocytic Leukaemia
Acronym: HIT-CLL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Collaborators: American Society of Hematology (Other)
Responsible Party: Principal Investigator, David Bartlett, Senior Lecturer, University of Surrey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FHMS 21-22 263 EGA
Record Dates: First submitted 2024-02-09; First posted 2024-04-23 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Chronic Lymphocytic Leukemia; Frailty; Muscle Function; Immune Function; Lipid Cell; Tumor
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Frailty; Neoplasms

STUDY DESIGN:
Intervention Model Description: Recruited participants will be randomised to either exercise only, exercise + nutritional guidance, or control for 12 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HIT Group (Experimental): Exercise Only
  * 3 sessions per week
  * Aerobic + Resistance Exercises
  Interventions: Behavioral: HIT
- EXE+ Group (Experimental): Exercise + Nutritional Guidance
  * 3 sessions per week
  * Aerobic + Resistance Exercises
  * Dietary assessment at baseline and during with guidance on eating a healthy diet provided
  Interventions: Behavioral: EXE+ Nutritional Guidance
- Control Group (No Intervention): Control group will receive no exercise or nutritional guidance

INTERVENTIONS:
Behavioral: HIT — Exercise training only
  Arms: HIT Group
Behavioral: EXE+ Nutritional Guidance — Exercise Training + Nutritional Guidance
  Arms: EXE+ Group

SUMMARY:
This randomised control clinical trial aims to investigate the effects of exercise training and diet on physical and functional fitness and immunological and metabolic changes in adults with chronic lymphocytic leukaemia. Investigators will randomise participants to either 12 weeks of supervised/semi-supervised exercise only, exercise + nutritional guidance, or no exercise.

DETAILED DESCRIPTION:
This study aims to perform a randomised control trial of exercise or exercise plus nutritional guidance on the physiological and immunological health of adults diagnosed with chronic lymphocytic leukaemia (CLL). Recruited participants will be randomised to either 12 weeks of an exercise-only program, an exercise-plus nutritional guidance program or a no-exercise control group. Fasting blood samples collected at Baseline and 12 weeks will measure absolute CLL cell counts, immune function, and inflammatory and metabolic biomarkers. A series of physical fitness assessments will be assessed at baseline and 12 weeks to determine physiologic reserve and resilience against external stressors. Additionally, participants will be asked to return 12 weeks after completing the intervention to assess the legacy effects of the intervention on the same physiological and blood-based biomarkers of health.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CLL (including small lymphocytic leukaemia) as per the International Workshop on CLL Guidelines.
* Male or female ≥ 18 years of age
* Able to walk on a treadmill or cycle on an ergometer
* Pass the Physical Activity Readiness Questionnaires (PAR-Q and PAR-Q+)

Exclusion Criteria:

* Corticosteroid therapy initiated less than 7 days before study entry. Prednisone 10mg or less or equivalent is allowed. Topical or inhaled corticosteroids are permitted.
* Secondary malignancy within 3 years of study enrollment requiring intervention except for adequately treated basal, squamous cell carcinoma or non-melanomatous skin cancer, carcinoma in situ of the cervix, superficial bladder cancer not treated with intravesical chemotherapy or BCG within 6 months, localised prostate cancer and PSA stable.
* Absolute contraindications to exercise: Recent (<6 months) acute cardiac event unstable angina, uncontrolled dysrhythmias causing symptoms or hemodynamic compromise, symptomatic aortic stenosis, uncontrolled symptomatic heart failure, acute pulmonary embolus, acute myocarditis or pericarditis, suspected or known dissecting aneurism and acute systemic infection.
* Significant orthopaedic limitations, musculoskeletal disease and/or injury. Due to the nature of the study, persons with known joint, muscle or other orthopaedic limitations that restrict physical activity may be excluded.
* Type I diabetes mellitus or uncontrolled Type II diabetes mellitus, or chronic obstructive pulmonary disease
* Uncontrolled blood pressure (≥180/90) at rest
* Known concurrent HIV, Hepatitis B or Hepatitis C
* Unable to comply with other study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2022-10-14 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in absolute number of CD19+/CD5+ CLL cells at week 12 | Baseline and 12 weeks
  A blood sample will be taken and assessed for CD19+/CD5+ CLL frequency using flow cytometry and total lymphocyte counts to determine the absolute number of CLL cells in x10^9/L
Change from baseline in cardiorespiratory fitness (CRF: VO2peak) at week 12 | Baseline and 12 weeks
  Cardiopulmonary exercise testing will be conducted to assess changes in fitness

SECONDARY OUTCOMES:
Frailty | Baseline and 12 weeks
  Frailty will be determined by a series of validated physical function tests that provide a score of 0-1(Robust), 2 (Pre-Frail), 3-5 (Frail)
Muscle Strength and Endurance | Baseline and 12 weeks
  Estimated one repetition maximum and repetitions to failure using machine-based weights
Muscle Health | Baseline and 12 weeks
  Ultrasound and near-infrared spectroscopy assessment of muscle fuel usage
Change in Quality of Life using the EORCT-QLQ-C30 | Baseline and 12 weeks
  Quality of life will be determined by the EORCT-QLQ-C30 questionnaire
Change in muscle oxygen metabolism during a single bout of exercise | Baseline and 12 weeks
  Measurement of muscle oxygenation via near infrared spectroscopy during a single session of acute exercise
Change in B-CLL Cell Function | Baseline and 12 weeks
  Measurement of in vitro B-CLL cell proliferation by flow cytometry
Change in systemic and cellular bioenergetics | Baseline and 12 weeks
  Measurement of in vitro immune cell fuel utilisation by high resolution respirometry and mass spectrometry

OTHER OUTCOMES:
Legacy Effect of Intervention on change in cardiorespiratory fitness (VO2peak) as measured by a cardiopulmonary exercise test | 12 weeks to 24 weeks
  Reassessment of CRF following 12 weeks of unguided exercise training
Legacy Effect of Intervention on absolute number of CD19+/CD5+ CLL cells | 12 weeks to 24 weeks
  Reassessment of absolute number of CD19+/CD5+ CLL cells following 12 weeks of unguided exercise training

CONTACTS AND LOCATIONS:
Overall Officials: David Bartlett, PhD, Principal Investigator — University of Surrey
Locations (1):
- University of Surrey, Guildford, United Kingdom

IPD SHARING:
Plan to Share IPD: No